CLINICAL TRIAL: NCT00159302
Title: A Pilot Study to Evaluate and Develop Biomarkers of iNOS Activity in Patients With COPD or Asthma and Healthy Volunteers
Brief Title: Biomarkers of iNOS Activity in COPD, Asthma, Healthy Control
Status: Withdrawn | Type: Observational
Why Stopped: Lead Researcher left the Department
Sponsor: Imperial College London (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: RES11115
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Healthy Smokers; Healthy Non-smokers; Patients With Mild Asthma; Patints With COPD (GOLD II)
MeSH Terms: interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

INTERVENTIONS:
Procedure: Induced Sputum
Procedure: Exhaled Nitric Oxide
Procedure: Nasal Nitric Oxide
Procedure: Blood Tests
Procedure: 24hr Urine Samples
Procedure: Exhaled Breath Condensate
Procedure: Spirometry

SUMMARY:
This pilot study will measure the baseline levels and the intra- and inter-subject variability of exhaled (alveolar and bronchial) and nasal NO in smoking subjects with mild and moderate COPD on or off steroid treatment, smoking healthy volunteers and non-smoking mild asthmatics off steroids, using multiple exhalation flow rates.

I

DETAILED DESCRIPTION:
n addition, exploratory markers of iNOS activity (eg. 3-nitrotyrosine, nitrite, nitrate and 3-nitro-4-hydoxyphenylacetic acid) in blood, sputum, urine and exhaled breath condensate will be evaluated. We will also evaluate exhaled and nasal NO in a population of mild asthmatics in order to obtain baseline and variability data for future clinical studies involving asthmatic subjects.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers (smokers)

1. Healthy subjects, defined as individuals who are free from significant cardiac, pulmonary, gastrointestinal, hepatic, renal, haematological, malignancy, endocrine, neurological and psychiatric disease as determined by history, physical examination and screening investigations.
2. Aged 40-75 years inclusive.
3. Male or female
4. Body mass index within the range 19-32kg/m2 inclusive.
5. Subject has a screening FEV1 measurement of > 80% of predicted
6. Capable of giving informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
7. Smokers with a pack history >10 pack years [number of pack years = (number of cigarettes per day / 20) x number of years smoked].

A smoking COPD subject will be eligible for inclusion in this study only if all of the following criteria apply:

1. COPD patients, defined as either Stage I or Stage II COPD diagnosis according to GOLD criteria Individuals must be otherwise healthy, individuals who are free from significant cardiac, gastrointestinal, hepatic, renal, haematological, malignancy, endocrine, neurological and psychiatric disease as determined by history, physical examination and screening investigations.
2. Aged 40-75 years inclusive.
3. Male or female
4. Body mass index within the range 19-32kg/m2 inclusive.
5. FEV1/FVC < 70%
6. FEV1 <15% reversibility (not % predicted) or an increase of <200ml (or both) after inhaled B2-agonists (400mcg salbutamol)
7. Capable of giving informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

9. An active smoker with a pack history of >10 pack years [number of pack years = (number of cigarettes per day / 20) x number of years smoked].

Asthma (non-smokers)

1. Individuals must be otherwise healthy, individuals who are free from significant cardiac, gastrointestinal, hepatic, renal, haematological, malignancy, endocrine, neurological and psychiatric disease as determined by history, physical examination and screening investigations.
2. Male or female
3. Body mass index within the range 19-32kg/m2 inclusive.
4. Capable of giving informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
5. Subjects with a history of non-severe allergic asthma and who are not receiving treatment in the form of inhaled or oral corticosteroids. Their history of asthma must be documented for a minimum of 6 months prior to entry to the study, with exclusion of other significant pulmonary diseases (i.e. chronic bronchitis, emphysema, bronchiectasis, cystic fibrosis, and bronchopulmonary dysplasia).
6. Aged 18 45 years
7. Baseline FEV1 > 70% of predicted
8. Non Smokers with no smoking history
9. PC20 methacholine < 8 mg/ml at screening
10. Subjects must have had positive skin prick test for 2 or more of common antigens in the past 2 years or at screening

Exclusion Criteria:

Healthy volunteers (smokers)

A healthy smoking subject will not be eligible for inclusion in this study if any of the following criteria apply:

1. As a result of the medical interview, physical examination or screening investigations, the Physician Responsible considers the volunteer unfit for the study.
2. The subject has participated in a study with a new molecular entity during the previous 4 months or any other clinical trial during the previous 3 months. In case of a non invasive, clinical trial not involving new molecular entities a 1 month washout will be sufficient.
3. The subject has donated a unit of blood within the previous month or intends to donate in the month after completing the study
4. The subject regularly, or on average, drinks more than 21 units per week
5. The subjects is taking any medication (whether prescribed or over-the-counter), any herbal medication (incl. St.John's Wort) or high doses of nutritional supplements which could interfere with the study tests, within 14 days of study entry and throughout the study.
6. The subject has received oral steroids within 3 months of study entry
7. The subject significant risk factors for Hepatitis B or C infection
8. The subject has significant risk factors for HIV infection.

COPD (smokers)

A smoking COPD subject will not be eligible for inclusion in this study if any of the following criteria apply:

1. As a result of the medical interview, physical examination or screening investigations, the Physician Responsible considers the volunteer unfit for the study.
2. The subject has participated in a study with a new molecular entity during the previous 4 months or any other clinical drug trial during the previous 3 months. In case of a non invasive, clinical trial not involving new molecular entities a 1 month washout will be sufficient.
3. The subject has donated a unit of blood within the previous month or intends to donate in the month after completing the study
4. The subject regularly, or on average, drinks more than 21 units per week
5. The subjects is taking any medication (whether prescribed or over-the-counter), any herbal medication (incl. St.John's Wort) or high doses of nutritional supplements which could interfere with the study tests, within 14 days of study entry and throughout the study.
6. The subject has received oral steroids within 3 months of study entry.
7. The subject has history of an upper respiratory infection (including sinusitis) within 4 weeks prior to study entry.
8. The subject has been hospitalised for a COPD exacerbation within 3 months of study entry
9. Subject is unable to abstain from xanthines (theophylline), inhaled long acting beta-2 agonists and tiotropium from 4 hours prior to first study visit until completion of study visit
10. For the non-steroid group, inhaled steroid use is not permitted within 14 days of study entry until completion of the study
11. The subject significant risk factors for Hepatitis B or C infection
12. The subject has significant risk factors for HIV infection. Asthma (non-smokers)

A non smoking asthmatic subject will not be eligible for inclusion in this study if any of the following criteria apply:

1. The subject has a history of life-threatening asthma, defined as an asthma episode that required intubation and/or was associated with either hypercapnoea, respiratory arrest or hypoxia seizures.
2. Subjects have a symptomatic pattern suggestive of poorly controlled asthma that in the opinion of the investigator precludes them from entry into the study
3. The subject received inhaled steroid within 14 days of study entry. Any subject who needs inhaled, intranasal or topical steroids between screening and study start should not be included in the study.
4. As a result of the medical interview, physical examination or screening investigations, the Physician Responsible considers the volunteer unfit for the study.
5. The subject has participated in a study with a new molecular entity during the previous 4 months or any other clinical drug trial during the previous 3 months. In case of a non invasive, clinical trial not involving new molecular entities a 1 month washout will be sufficient.
6. The subject has donated a unit of blood within the previous month or intends to donate in the month after completing the study
7. The subject regularly, or on average, drinks more than 21 units per week
8. The subjects is taking any medication (whether prescribed or over-the-counter), any herbal medication (incl. St.John's Wort) or high doses of nutritional supplements which could interfere with the study tests, within 14 days of study entry and throughout the study.
9. The subject has received oral steroids within 3 months of study entry
10. The subject has history of a respiratory infection (including sinusitis) within 4 weeks prior to study entry
11. The subject has been hospitalised for a asthma exacerbation within 3 months of study entry
12. The subject has tested positive for hepatitis C antibody or hepatitis B surface antigen or a positive medical history for hepatitis C antibody or hepatitis B surface antigen.
13. History of current or past drug or alcohol abuse.
14. Subject is unable to abstain from xanthines (theophylline), inhaled long acting beta-2 agonists and tiotropium from 4 hours prior to first study visit until completion of study visit.
15. Current or past smoking history.
16. The subject significant risk factors for Hepatitis B or C infection
17. The subject has significant risk factors for HIV infection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2003-09 (Actual); Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sergei A Kharitonov, MD PhD, Principal Investigator — Imperial College London
Locations (1):
- Section of Airway Disease, Asthma Lab, Imperial College London, Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No